CLINICAL TRIAL: NCT06646198
Title: Transjugular Intrahepatic Portosystemic Shunt (TIPS) Plus Half-dose Donafenib (a Kind of Anti-angiogenesis Agents) in Advanced HCC with Tumor Thrombosis-associated Portal Hypertension: a Prospective, Single-arm, Phase II Study. (DoTH Study)
Brief Title: TIPS Plus Half-dose Donafenib in AHCC with PVTT-associated Portal Hypertension
Acronym: DoTH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fei Gao (Other)
Responsible Party: Sponsor-Investigator, Fei Gao, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DoTH
Record Dates: First submitted 2024-10-14; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma with PVTT
Keywords: Transjugular intrahepatic portosystemic shunt (TIPS); Hepatocelluar Carcinoma with portal vein tumor thrombus; tumor thrombosis-associated portal hypertension; Donafenib; Combination therapy
MeSH Terms: interventions — Portasystemic Shunt, Transjugular Intrahepatic; donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DoTH: TIPS plus half-dose donafenib (Experimental): TIPS plus half-dose donafenib
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt (TIPS); Drug: Donafenib

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt (TIPS) — Perform transjugular intrahepatic portosystemic shunt under the guidance of DSA
Drug: Donafenib — Half-dose donafenib, 100mg BID P.O. unless any evidence of disease progression or unacceptable side effects.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of transjugular intrahepatic portosystemic shunt (TIPS) plus half-dose donafenib (a kind of anti-angiogenesis agents) in advanced hepatocellular carcinoma (BCLC-C Stage) accompanied by tumor thrombosis-associated portal hypertension.

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase II study to evaluate the efficacy and safety of transjugular intrahepatic portosystemic shunt (TIPS) plus half-dose donafenib (a kind of anti-angiogenesis agents) in advanced hepatocellular carcinoma (BCLC-C Stage) accompanied by tumor thrombosis-associated portal hypertension. Subjects who meet the admission criteria will be treated with half-dose donafenib after TIPS until disease progression, intolerable toxicity, death, withdrawal of the patient, or the researchers determined that the drug must be discontinued.

The primary outcome measure is to evaluate the objective response rate (ORR) based on mRECIST. The secondary outcome measures include the duration of response (DOR), disease control rate (DCR), the recurrence rate of portal hypertension-related haemorrhage or ascites, the median progression-free survival time (mPFS) and median overall survival time (mOS). This study also aims to assess the safety and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joined the study and signed an informed consent form;
2. ≥18 and ≤ 75 years old, both male and female;
3. Pathologically confirmed hepatocellular carcinoma, at least one measurable focus without local treatment (according to mRECIST or RECIST 1.1 requirements;
4. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1
5. BCLC-C stage accompanied by tumor thrombosis-associated portal hypertension;
6. Newly diagnosed patients who have not received local or systemic therapy in the past;
7. Expected survival period ≥ 3 months;
8. The functions of vital organs meet the following requirements (no blood components, cell growth factors and other corrective treatment drugs are allowed within 14 days before the first administration): the absolute count of neutrophils≥1.5×10^9/L; Platelet ≥50×10^9/L; Hemoglobin ≥60 g/L; Serum albumin ≥28 g/L; Thyroid-stimulating hormone (TSH)≤1×ULN (if abnormal, the levels of FT3 and FT4 should be examined at the same time, if the levels of FT3 and FT4 are normal, they can be included in the group); Bilirubin≤2×ULN (within 7 days before the first administration); ALT and AST ≤5×ULN (within 7 days before the first dose); Serum creatinine≤1.5×ULN;
9. Child-Pugh score ≤ 13 points;
10. Diagnosed with portal hypertension-related complications: Gastrointestinal bleeding; refractory or recurrent ascites; hepatic pleural effusion; portal vein tumor thrombus exceeds 50% of lumen area.
11. Non-surgical sterilization or female patients of childbearing age need to use a medically approved contraceptive method (such as an intrauterine device, contraceptive, or condom) during the study treatment period and within 3 months after the end of the study treatment period; Female patients of childbearing age who undergo surgical sterilization must be negative in serum or urine HCG within 72 hours before enrollment in the study; and must be non-lactating; for male patients whose partners are women of childbearing age, at the last time use effective methods for contraception within 3 months.

Exclusion Criteria:

1. The patient has any active autoimmune disease or a history of autoimmune disease;
2. The patient is using immunosuppressive agents or systemic hormone therapy to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other curative hormones), and continues to use it within 2 weeks before enrollment;
3. Severe allergic reaction to any compositions of donafenib tablets or contrast media containing iodine ;
4. Central nervous system metastasis;
5. Patients who have received liver transplantation in the past;
6. Tumor thrombus beyond the portal vein range, such as hepatic vein, inferior vena cava, right atrium, splenic vein, superior mesenteric vein;
7. Suffer from high blood pressure and cannot be well controlled by anti-hypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
8. Uncontrolled cardiac clinical symptoms or diseases, such as: NYHA level 2 or higher heart failure, unstable angina pectoris, myocardial infarction occurred within 1 year, clinically significant supraventricular or ventricular arrhythmia requires treatment or intervention , QTc>450ms (male); QTc>470ms (female); Abnormal coagulation function (INR>2.0, PT>16s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy, and allow the preventive use of low-dose aspirin and low molecular heparin;
9. Child-Pugh score >13 points;
10. Arterial/venous thrombosis events that occurred within 6 months before randomization, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
11. Known genetic or acquired bleeding and thrombotic tendency (such as hemophilia patients, coagulation dysfunction, thrombocytopenia, etc.);
12. Urine routine test showed urine protein ≥ ++ and confirmed 24-hour urine protein content> 1.0 g;
13. The patient has active infection, fever of unknown origin within 7 days before medication ≥38.5℃, or baseline white blood cell count >15×109/L;
14. Patients with congenital or acquired immune deficiencies (such as HIV-infected persons);
15. Moderate to severe pulmonary hypertension, pulmonary artery pressure was assessed by ultrasound >40mmHg；
16. The patient suffered from other malignant tumors in the past 3 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ);
17. The patient has previously received other anti-PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or has previously received apatinib therapy;
18. According to the judgment of the investigator, the patient has other factors that may affect the results of the study or cause the study to be terminated halfway, such as alcoholism, drug abuse, other serious diseases (including mental illness) that require combined treatment, and other abnormalities which may affect the efficacy and/or safety of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 and mRECIST | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to 1 year)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1 or mRECIST

SECONDARY OUTCOMES:
Overall survival (OS) | From the start date of the TIPS until date of death from any cause, assessed up to 2 years.
  OS is measured from the start date of the TIPS until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes earlier, assessed up to 2 years.
Progression-free survival (PFS) | The progression-free survival (PFS) defined as the time from the date of TIPS to the date of first documented progression (mRECIST or RECIST v1.1) or date of death from any cause, whichever came first, assessed up to 2 years
  The progression-free survival (PFS) defined as the time from the date of TIPS to the date of first documented progression (mRECIST or RECIST v1.1) or date of death from any cause, whichever came first, assessed up to 2 years
Disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to 1 year)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1 or mRECIST.
Rate of portosystemic shunt stent patency | 1, 3, 6, 9, 12 months after TIPS
  The status of the shunt stent evaluated by the color Doppler ultrasound.
Recurrence rate of portal hypertension-related complications | From date of TIPS until portal hypertension-related complications (up to 6 months)
  It was defined as the percentage of patients with recurrent gastrointestinal bleeding, refractory ascites, hepatic pleural effusion, and portal hypertensive gastroenteropathy within 6 months after TIPS

OTHER OUTCOMES:
Treatment-related adverse events | From the start date of the Treatment Phase until date of death from any cause (up to 1 year)
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Gao, M.D.，Ph.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No